CLINICAL TRIAL: NCT01072084
Title: Endomicroscopy in Patients With Food Allergy: a New Diagnostic Option
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, yurdagül zopf, Professor Dr., University of Erlangen-Nürnberg Medical School
Other Study IDs: FAEM
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Food Allergy
Keywords: food allergy; confocal laser endoscope; diagnosis; Diagnosis of food allergy
MeSH Terms: conditions — Food Hypersensitivity; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with food allergy
- Healthy subjects

SUMMARY:
The purpose of this study is to evaluate the endoscopic diagnostic options of the endomicroscopy in patients with food intolerance.

DETAILED DESCRIPTION:
Food allergy is with a prevalence of 2-4% a seldom disease. The endoscopy of the gastrointestinal tract and the histological analysis of taken biopsies of the intestinal mucosa are basic instruments in the diagnostic of food allergy. With modern high-resolution video endoscopy the intestinal mucosa can be investigated on inflamed areas and can evaluate several of differential diagnosis. With the implementation of a fluorescein based confocal laser endoscope the intestinal mucosa can be magnified 1000 fold, so that even next to the macroscopic investigation the cellular patterns can be analyzed. The laser endoscope offers for the first time an in vivo presentation of cellular structures. Our study group could utilise for the first time the laser endoscope in patients with colitis ulcerosa for cancer prevention. Hereby, the cancer prediction could be enhanced obviously. Furthermore, we conducted these investigations in more than 1500 patients und could present that this method is a safety method.

Based on these investigations we want to implement now the laser endoscope in the diagnostic field of food allergy. Patient wit food allergy generates through the intestinal mediators and histamine secretion an oedema, an increase of inflammatory cells, vasodilatation and expansion of lymph nodes. In comparison of patients with food allergy to healthy subjects, the degree of oedema formation, the amount of cell infiltration and the expansion of lymph nodes will be evaluated.

The aim of the present study is to detect these cellular structures in patients with food allergy and to open with that a new diagnostic option in patient with an allergy disease.

ELIGIBILITY:
Inclusion Criteria:

* new diagnosed and not treated patients with food allergy

Exclusion Criteria:

* decreased clotting (Quick < 50%, platelet < 50.000/µl)
* not given consent
* known allergy against fluorescein
* pregnant and breastfeeding woman

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both study groups will be acquired from the ambulant gastrointestinal consultation of the Medical department 1 of the Universityhospital Erlangen.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The degree of oedema formation, the amount of cell infiltration and the expansion of lymph nodes. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Raithel, MD, Principal Investigator — Medical Department 1, University hospital Erlangen
Locations (1):
- Medical Department 1, University hospital Erlangen, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Kiesslich R, Goetz M, Lammersdorf K, Schneider C, Burg J, Stolte M, Vieth M, Nafe B, Galle PR, Neurath MF. Chromoscopy-guided endomicroscopy increases the diagnostic yield of intraepithelial neoplasia in ulcerative colitis. Gastroenterology. 2007 Mar;132(3):874-82. doi: 10.1053/j.gastro.2007.01.048. Epub 2007 Jan 31. PMID 17383417